CLINICAL TRIAL: NCT03431155
Title: The Impact of Nursing Interventions Based on Uncertainty In Illness Theory on Uncertainty, Hopelessness, Coping And Adaptation for Care Givers Of Children With Cancer
Brief Title: The Impact of Nursing Interventions Based on Uncertainty In Illness Theory on Care Givers Of Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Sevil Özkan, Research Assistant, Nursing, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017/44
Record Dates: First submitted 2018-01-23; First posted 2018-02-13 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Pediatric Cancer; Nurse's Role
Keywords: children; cancer; care giver; uncertainty; nursing intervention; education
MeSH Terms: conditions — Neoplasms | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: * Data were collected by a nurse (not researher) who did not know anything about participants of experiment and control group.
  * Data recorded on the computer by another nurse (without specifying the experiment and control group)
  * The experimental and control groups codified by the co-investigator.
  * The analysis of the data encoded by the groups was done by a statistical expert. Data collectors, statistical analyzes and report writing were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Nursing intervention
  Interventions: Other: Nursing intervention
- Control Group (No Intervention): - Receive routine nursing care

INTERVENTIONS:
Other: Nursing intervention — Nursing Intervention: Protocol and education booklet were developed according to literature and Theory. There were six modules (10 session) which aimed to personal education for every care givers. Every session took 20 minutes and total 200 minutes. First 5 modules finished within 3 days and aafter one week last module completed (to summarize process). Also individual counseling were made.
  Arms: Experimental group

SUMMARY:
The aim of this Randomised Controlled study was to determine the effect of nursing interventions based on Mishel's Uncertainty in Illness Theory on uncertainty, hopelessness, coping and compliance for care givers' of children with cancer. Sample was 46 (experimental group:23; control group: 23) cara givers of children. Experimental group received nursing interventions (6 modules, 200 minutes nursing education) based on Mishel's Uncertainty in Illness Theory while control group received routine hospital care. Data were collected 3 times: pre test, post test (2 weeks after intervention for experimental group or two weeks after from pretest for control group), and follow up (2 weeks after post tests).

DETAILED DESCRIPTION:
Cancer defines a group of diseases that arise from the uncontrolled proliferation and spread of abnormal cells. The prevalence of cancer before the age of 15 years is 110-150 million. Every year, more than 150,000 people in the World are newly diagnosed, and over 10,000 children in America are diagnosed with cancer for the first time. It is reported that 2500-3000 new cases of childhood cancer are expected to be seen in our country, Turkey, annually.

Childhood cancer is a major stressor for family. They are at risk for developing psychosocial problems during the course of disease and its long and stressful treatment. And uncertainty is one of these problems which they live. Uncertainty arises when "the decision maker can not give a definite value to a certain event or situation" or "can not predict the accuracy of the results". Uncertainty refers to the inability to identify, interpret and predict the disease-related condition/event. Uncertainty can have positive or negative affects to child and family according the meaning and coping of uncertainty.

Mishel is the first nurse theorist who mentioned uncertainty in illness in the aspect of nursing as a theory. In her theory, nursing interventions can help care giver to cope with or adapt the uncertainty. Nursing interventions should contain the main domains of such as communication, education, supporting, being reliable health care professional for parents.

In this study, 46 care givers of children with cancer from two different university hospitals in Turkey. They were assigned group by using closed envelops that contain the letter of E(experimental) or C(control). Prior to study, sample size for each group calculated according to effect size (d=0,20), power (.80), alfa error (.05) and it was found 42 for all group. To avoid possible sample problems can be seen during to study (such as do not want to continue the stud etc), sample was improved %10 and sample number were decided 46 care giver in total. During the study while 18 care giver (9 from experimental, 9 from control group) finished the study, we calculated real effect size of our study and it was foun 0.24 and according to it we calculated sample size again and it was 30 in total. So we decided to continiue our study with 46 participants.

Experimental group received nursing intervention according to protocol. It contained 6 modules (total 10 personal education session) that were developed based on Theory and literature. The aim of this intervention was to control/solve the antecedents of uncertainty and to affect appraisal of uncertainty in a positive way so care givers could improve the coping and adaptation of uncertainty. Control group received routine nursing intervention that was given normally for hospitals to avoid bias and ethical problems.

Data was collected using information form (information about participant, parents and children), three scales (Turkish Version of Parents' Perception Uncertainty in Illness Scale: Parent/Child Form, Beck's Hopelessness Scale, Coping and Adaptation Process Scale). Scales validation and reliability studies were made for Turkish population.

ELIGIBILITY:
Inclusion criteria:

* Care giver of children with cancer who is next to children during the hospital process.
* Children diagnosed and continued to clinical therapy in one of two university hospitals.
* At least have the primary education (5 year education)
* Child get at least one cure chemotherapy/radiotherapy
* Care givers' age must be et least 18 year-old
* Care giver can speak and understand Turkish fluently

Exclusion Criteria:

* Care giver with psychiatric disorder
* Child has loss of function due to cancer related operation (amputation, etc)
* Having a child whose treatment of cancer finished
* Having a child whose disease is in remission
* Having a child whose disease relapse
* Having a child who is terminal term
* Having a child who is older than 18 year-old
* Prior to cancer diagnosis, children have a dhronic disease or genetic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Less uncertainty | At the end of 4 week.
  Means of Parents Perceived Uncertainty in Illness Scale: Parent/child From for participants in experimental group will be less.

SECONDARY OUTCOMES:
Less hopelessness | At the end of 4 week.
  Means of Beck Hopelessness Scale for participants in experimental group will be less.
More coping and adaptation | At the end of 4 week.
  Means of Coping and Adaptation Processing Scale for participants in experimental group will be more.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not plan to share any data of participants.